CLINICAL TRIAL: NCT06803485
Title: Effect of Venlafaxine Versus Dosulepin on Clinical Outcomes, Neuroinflammation and Cortisol Level in Pain Predominant Somatic Symptom Disorder: A Group-sequential Randomized Controlled Trial
Brief Title: Effect of Venlafaxine Versus Dosulepin in Pain Predominant Somatic Symptom Disorder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGThesis/2024-25/108
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Somatic Symptom Disorder (DSM-V)
Keywords: Somatic symptom disorder; Dosulepin; Venlafaxine; Somatic syndrome disorder with pain predominance; Cortisol; TNF alpha
MeSH Terms: interventions — Venlafaxine Hydrochloride; Dothiepin

STUDY DESIGN:
Intervention Model Description: Group Sequential Study Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venlafaxine group (Experimental): Venlafaxine will be started at dose of 37.5mg/day in first week and increased to a stable dose of 75 mg/day from second week and will be continued till 8 weeks.
  Interventions: Drug: Venlafaxine
- Dosulepin group (Active Comparator): Dosulepin will be started at dose of 25 mg/day in first week and increased to a stable dose of 50 mg/day from second week and will be continued till 8 weeks.
  Interventions: Drug: Dosulepin

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxine will be started at a dose of 37.5 mg/day in first week and increased to a stable dose of 75 mg/day from second week and will be continued till 8 weeks.
  Arms: Venlafaxine group
Drug: Dosulepin — Dosulepin will be started at a dose of 25 mg/day in first week and increased to a stable dose of 50 mg/day from second week and will be continued till 8 weeeks.
  Arms: Dosulepin group

SUMMARY:
Somatic symptom disorder (SSD) is marked by persistent physical complaints, often involving pain, alongside excessive thoughts or behaviors related to health, which substantially disrupt daily functioning. The underlying mechanisms of SSD are multifaceted. The serotonin hypothesis links low serotonin levels to the development of somatic symptoms, while the cortisol hypothesis highlights dysregulation of the hypothalamic-pituitary-adrenal (HPA) axis, with chronic stress often associated with hypocortisolism. Furthermore, the neuroinflammatory hypothesis suggests that cytokine-driven inflammation and activation of glial cells may intensify pain and somatic symptoms, exacerbating patient outcomes. Challenges such as limited acceptance of the diagnosis, resistance to treatment among patients and caregivers, and societal stigma further hinder effective management.

Currently, treatment options lack definitive efficacy, with pharmacological interventions primarily targeting serotonin pathways. There is limited exploration of therapies addressing mechanisms like cortisol dysregulation and neuroinflammation. Commonly used medications include tricyclic antidepressants (TCAs), serotonin-norepinephrine reuptake inhibitors (SNRIs), and selective serotonin reuptake inhibitors (SSRIs), with prescribing decisions often based on physician discretion and patient tolerance rather than clear evidence favoring one class over another.

The proposed study aims to compare the efficacy and safety of Dosulepin (a TCA) and Venlafaxine (an SNRI) in managing SSD patients with predominant pain. By evaluating their impact on symptom severity, quality of life, and biomarkers such as serum cortisol and TNF-alpha levels, this research seeks to enhance understanding of SSD treatment. The findings aim to address gaps in SSD pharmacotherapy and contribute to improved patient care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of somatic symptom disorder with pain predominance (DSM-5).
* Patients of either sex within the age group of 18-65 years.
* Patients with PHQ-15 score of ≥ 5.
* All included patients will be treatment-naïve or have not received any treatment in the last 4 weeks.
* Patients who have given written informed consent.

Exclusion Criteria:

* A diagnosed psychological condition that might require other treatment (e.g., psychosis, suicidality)
* Patient undergoing current psychotherapy.
* Patients with cognitive impairment.
* History of allergy to either of the study drugs (dosulepin or venlafaxine).
* Patients with comorbidities like any malignancies, hepatic, renal, cardiovascular, neurological or endocrinal, or respiratory dysfunction.
* Substance abuse history of psychoactive agents.
* Pregnant and lactating mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of Somatic Symptom Disorder using PHQ-15 (Patient health questionnaire) score | 8 weeks
  The PHQ-15 is a freely accessible self-administered somatic symptoms scale that is based on the full Patient Health Questionnaire. Screening for 15 somatic symptoms.Each symptom is scored as 0, 1, or 2, with the total score ranging from 0 to 30. The scores of <5, 5-9, 10-14, and 15-30 indicate minimal, low, moderate, and high symptom levels, respectively.

SECONDARY OUTCOMES:
Treatment response rate | 8 weeks
  Treatment response rate (defined as a reduction of ≥ 50% of the PHQ-15 score from baseline) will be evaluated.
Change in serum cortisol | 8 weeks
  Change in serum levels of cortisol at baseline after 8 weeks from baseline will be evaluated.The sample will be collected at 8 am.
Change in serum Tumor necrosis factor (TNF) alpha levels | 8 weeks
  Change in serum levels of TNF-α after 8 weeks from baseline will be evaluated.
Change in quality of life | 8 weeks
  Quality of life will be evaluated using WHO-QOL BREF scores after 8 weeks from baseline. A condensed version of the WHOQOL-100 questionnaire, the WHOQOL-BREF has 26 items. There are four domains, namely, Physical (domain 1), Psychological (domain 2), Social (domain 3), and Environmental (domain 4) in WHOQOL-BREF. Each question will be evaluated on a scale of 1-5. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
Incidence of treatment-emergent adverse events | 8 weeks
  The Antidepressant Side-Effect Checklist (ASEC) will be used to evaluate the incidence of adverse events. 21 symptom-specific questions are evaluated on a 0-3 scale with "0" denoting absence, "1" denoting mild, "2" denoting moderate, "3" denoting severe, the final score lies in the range of 0-63. Additionally, the scale determines whether a symptom is associated with antidepressants.

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study will be shared with qualified researchers upon reasonable request. Data will be available after publication and subject to review of a data access proposal and data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication of data and will be for next 5 years.
Access Criteria: Data will be shared with qualified researchers upon reasonable request and subject to review of a data access proposal and data use agreement.

REFERENCES:
- [Background] Miyauchi T, Tokura T, Kimura H, Ito M, Umemura E, Sato Boku A, Nagashima W, Tonoike T, Yamamoto Y, Saito K, Kurita K, Ozaki N. Effect of antidepressant treatment on plasma levels of neuroinflammation-associated molecules in patients with somatic symptom disorder with predominant pain around the orofacial region. Hum Psychopharmacol. 2019 Jul;34(4):e2698. doi: 10.1002/hup.2698. Epub 2019 May 24. PMID 31125145
- [Background] Park B, Lee S, Jang Y, Park HY. Affective dysfunction mediates the link between neuroimmune markers and the default mode network functional connectivity, and the somatic symptoms in somatic symptom disorder. Brain Behav Immun. 2024 May;118:90-100. doi: 10.1016/j.bbi.2024.02.017. Epub 2024 Feb 13. PMID 38360374
- [Background] Rief W, Auer C. Cortisol and somatization. Biol Psychol. 2000 May;53(1):13-23. doi: 10.1016/s0301-0511(00)00042-9. PMID 10876062
- [Background] Kurlansik SL, Maffei MS. Somatic Symptom Disorder. Am Fam Physician. 2016 Jan 1;93(1):49-54. PMID 26760840
- [Background] D'Souza RS, Hooten WM. Somatic Symptom Disorder. 2023 Mar 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532253/ PMID 30335286
- [Background] Toussaint A, Kroenke K, Baye F, Lourens S. Comparing the Patient Health Questionnaire - 15 and the Somatic Symptom Scale - 8 as measures of somatic symptom burden. J Psychosom Res. 2017 Oct;101:44-50. doi: 10.1016/j.jpsychores.2017.08.002. Epub 2017 Aug 2. PMID 28867423